CLINICAL TRIAL: NCT04901754
Title: Camrelizumab Plus Apatinib as Maintenance Treatment in Extensive-stage SCLC With a Response or Stable Disease After Standard Chemotherapy: A Single-arm, Prospective Clinical Trial
Brief Title: Camrelizumab Plus Apatinib as Maintenance Therapy in Extensive-stage Small-cell Lung Cancer
Acronym: CAMERA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA-SCLC-Ⅱ-002
Record Dates: First submitted 2021-05-20; First posted 2021-05-25 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-03

CONDITIONS: Small Cell Lung Carcinoma
Keywords: Maintenance; Camrelizumab Plus Apatinib
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — camrelizumab; apatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Camrelizumab Plus Apatinib (Experimental): camrelizumab 200 mg administered intravenously (IV) on Day 1 of each 21-day cycle plus Apatinib capsules 250 mg given orally
  Interventions: Drug: Camrelizumab Plus Apatinib

INTERVENTIONS:
Drug: Camrelizumab Plus Apatinib — -Drug: camrelizumab Camrelizumab intravenous infusion was administered at a dose of 200 mg on Day 1 of each 21-day cycle,until PD.
  Other Name: SHR-1210
  -Drug: Apatinib Mesylate Apatinib capsules 250 mg given orally , once daily in 21-day cycle ,until PD.

SUMMARY:
This single-arm, Phase II study was designed to evaluate the safety and efficacy of Camrelizumab (anti-programmed death-receptor 1 [PD-1] antibody) combination with Apatinib in participants with ES-SCLC who was response or stable disease after firstline standard chemotherapy. Participants will be receive camrelizumab +apatinib on 21-day cycles until progressive disease (PD) as assessed by the investigator using Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1). Treatment can be continued until persistent radiographic PD or symptomatic deterioration.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged 18 and 75 years old;
* Signed the informed consent form prior to patient entry;
* Eastern Cooperative Oncology Group performance status of 0 or 1;
* Expected Survival Time: Over 3 months;
* Pathological or cytologically proven extensive-Stage small cell lung cancer(according to Veterans Administration Lung Study Group)and without progression after Cycles 4-6 21-day cycles of first-line Standard chemotherapy(Evaluation was CR /PR/SD based on RECIST1.1);
* If prophylactic cranial irradiation (PCI) was not planned,informed consent was required to be written between 3 weeks and 5 weeks after day 1 of the last cycle of chemotherapy. If PCI was planned or already performe, informed consent was required to be written between 3 weeks and 8 weeks after day 1 of the last cycle of chemotherapy.

Exclusion Criteria:

* Has prior therapy with anti-programmed cell death (PD)-1, anti-PD-L1,anti Cytotoxic T lymphocyte-associated Antigen(CTLA)-4 or other Drugs that target T cells;
* Has prior therapy with angiogenesis inhibitors,Such as sunitinib, bevacizumab, apatinib, anlotinib;
* Has active or untreated central nervous system (CNS) metastases and/or cancerous meningitis;
* Imaging (CT or MRI) shows that tumor invades large blood vessels or the boundary with blood vessels is unclear;
* Has spinal cord compression which was not cured or relieved through surgery and/or radiotherapy, or diagnosed spinal cord compression after treatment showed no clinical evidence of disease stabilization prior to allocation ≥1 week;
* Within the past 2 weeks have used high dose antibiotics;
* According to the judgement of the researchers, there are other factors that may lead to the termination of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2021-07-14 (Actual); Primary Completion 2022-08-15 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Progression free survival(PFS) | up to 12 months
  From the date of maintenance randomization to the date of first document of progression or symptomatic deterioration, or death due to any cause

SECONDARY OUTCOMES:
Overall survival(OS) | up to 24 months
  From the date of maintenance randomization until death from any cause, with participants last known to be alive censored at the date of last contact

OTHER OUTCOMES:
Adverse events (AEs) | up to 24 month
  All adverse event/Serious adverse event that occurred during the study period according to CTCAE v 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Qiming Wang, Doctor, Principal Investigator — Henan Cancer Hospital
Locations (1):
- Henan Cancer Hospital, Zhengzhou, Henan, China